CLINICAL TRIAL: NCT04213313
Title: Consecutive, Case Control Study of Association Between Single Nucleotide Polymorphism of SP-D and Susceptibility and Prognosis of Infectious Keratitis
Brief Title: Association Between SNP of SP-D and Susceptibility and Prognosis of Infectious Keratitis
Acronym: ABSOSASAPOIK
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: IR2019001224; 2019-309 (Other Grant/Funding Number: 2nd Affiliated Hospital, School of Medicine, Zhejiang University)
Record Dates: First submitted 2019-12-24; First posted 2019-12-30 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2019-12

CONDITIONS: Infectious Keratitis
Keywords: Infectious Keratitis; surfactant protein D; single nucleotide polymorphisms; Met11Thr; rs721917
MeSH Terms: interventions — Base Sequence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — 6ml peripheral venous blood in healthy control populations and in patients with infectious keratitis.
  ulcerated marginal tissue in patients with infectious keratitis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: health volunteers
  Interventions: Other: Sequencing
- Infectious Keratitis Group: Infectious corneal patients
  Interventions: Drug: Treatment of bacterial keratitis; Drug: Treatment of fungal keratitis; Drug: Treatment of viral keratitis; Diagnostic Test: corneal scraping; Other: Sequencing

INTERVENTIONS:
Drug: Treatment of bacterial keratitis — 0.3% Levofloxacin Eye Drops or 0.3% Tobramycin Eye Drops QID
  Groups: Infectious Keratitis Group
Drug: Treatment of fungal keratitis — 1% Fluconazole Eye Drops or 0.25% Amphotericin B Eye Drops QID
  Groups: Infectious Keratitis Group
Drug: Treatment of viral keratitis — 0.1% Acyclovir eye drops QID ，Ganciclovir gel QN，Famiclovir tablets 0.25g TID
  Groups: Infectious Keratitis Group
Diagnostic Test: corneal scraping — culture and sensitivity of corneal ulcerated infiltrating edge tissue
  Groups: Infectious Keratitis Group
Other: Sequencing — polymerase chain reaction with sequence specific primers(PCR-SSP) and Sanger sequencing

SUMMARY:
This study explores the association between single nucleotide polymorphism (Met11Thr) of surfactant protein D(SP-D) and susceptibility and prognosis of infectious keratitis.Met11Thr of SP-D of patients with keratitis and normal controls were compared.Allele and genotype frequencies of patients with keratitis and normal controls were determined by polymerase chain reaction with sequence specific primers(PCR-SSPs) .SP-D gene polymorphism of patients with keratitis and normal controls was detected by Sanger sequencing

DETAILED DESCRIPTION:
Surfactant protein D(SP-D) plays an important role in the innate immune system of the eye in the lacrimal duct, cornea and conjunctiva.The single lipopolysaccharide on the surface of bacteria and the receptors on the surface of immune cells are linked by SP-D ,which acts as a bridge to neutralize viruses in the innate immune defense system and assists other immune cells in clearing bacteria and fungi.SP-D can also participate in the acquired immune response after combining with lipopolysaccharide on the surface of microorganisms.Some single nucleotide polymorphisms of SP - D can not only affect the plasma level of SP - D, which leads to the differences of pathogen defense capability, but also can affect the space configuration and structure of carbohydrate recognition domain of SP-D, causing the change of ability of SP - D combined with pathogens to influence its defensive role.The concentration of SP - D in ocular surface is closely related to the occurrence and progression of infectious keratitis.Association between single nucleotide polymorphisms of SP-D and the occurrence and development of infectious keratitis has yet to be confirmed by research.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Infectious Keratitis.
* Laboratory diagnosis of Infectious Keratitis.

Exclusion Criteria:

* Patients with topical or systemic long-term use of hormones, interferon, or immunosuppressive therapy.
* Patients with basic diseases such as diabetes, autoimmune disease, sjogren's syndrome, blepharitis, eyelid defect or incomplete eyelid closure.
* Patients with history of corneal myopia laser, cataract surgery and vitrectomy, or history of serious ocular trauma and drug allergies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with infectious keratitis at 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China between October 2016 to June 2019
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Base type | before the treatment
  Base type of SNP（rs721917）:(Met and Thr)
Genotype | before the treatment
  Genotype of SNP（rs721917）:( Met /Met , Thr/Thr and Met/Thr)

SECONDARY OUTCOMES:
Grading of Keratitis | before the treatment
  Grading of Keratitis：
  1. cornea:transparency ,edema,turbidity,perforation
  2. conjunctiva: hyperaemia
  3. blephar:inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Tao Jiang, Study Director — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Department of Ophthalmology, The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No